CLINICAL TRIAL: NCT06006793
Title: A Phase I, Dose-escalation/Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Anti-Tumor Activity of SY-5933 Tablets in Patients With Advanced KRAS p.G12C Mutant Solid Tumors
Brief Title: A Study of SY-5933 in Patients With Advanced Solid Tumors Harboring the KRAS p.G12C Mutation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shouyao Holdings (Beijing) Co. LTD (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SY-5933-I-01
Record Dates: First submitted 2023-08-10; First posted 2023-08-23 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Advanced Solid Tumor
Keywords: KRAS p.G12C Mutation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-escalation and Dose-expansion (Experimental): In dose-escalation phase, SY-5933 tablets will be administrated orally, repeat daily, 28 days as a dosing cycle, in ascending doses.
  In dose-expansion phase, RP2D of SY-5933 determined in dose-escalation phase will be administrated orally, repeat daily, 28 days as a dosing cycle.
  Interventions: Drug: SY-5933

INTERVENTIONS:
Drug: SY-5933 — KRAS p.G12C inhibitor
  Other Names: SY-5933 tablet

SUMMARY:
This is a single-arm, open-label, phase 1 study to evaluate the safety, tolerability, pharmacokinetics (PK), and anti-tumor activity of SY-5933 in patients with KRAS p.G12C mutant advanced solid tumors.

DETAILED DESCRIPTION:
The study will be conducted in 2 parts: Part 1 - Dose Escalation and Part 2 - Dose Expansion. Part 1 is aimed at evaluating the safety, tolerability, PK and pharmacodynamics of SY-5933 and determining the recommended phase II dose (RP2D) of repeat daily (QD) dosing schedule in subjects with advanced KRAS p.G12C mutant solid tumors using accelerated titration and 3+3 design. The dose escalation part of the study will consist of 7-13 subjects and the dose expansion part will consist of 30-60 additional subjects, comprising 2 cohorts. Cohort A includes patients with non-small cell lung cancer (NSCLC) harboring KRAS p.G12C mutations and Cohort B includes patients with other advanced solid tumors (colorectal, pancreatic cancers, etc.). Patients in dose expansion study will receive SY-5933 tablets QD, oral administration, 28 days as a dosing cycle, to further evaluate the safety, PK profile, and efficacy of SY-5933, and to further define RP2D. Administration of SY-5933 may continue until evidence of disease progression, intolerance to SY-5933, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 18 years old
2. Eastern Collaboration Oncology Group (ECOG) performance status (PS) scored of 0-1.
3. Estimated life expectancy >12 weeks.
4. Patients must have at least one assessable lesion in the dose-escalation part and one measurable lesion in the dose-expansion part per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
5. In the dose-escalation part, patients must have histologically or cytologically confirmed advanced solid tumors harboring the KRAS p.G12C mutation and have progressed after standard therapy, or standard therapy is inappropriate or unavailable.

   In the dose-expansion part, patients must have histologically or cytologically confirmed advanced KRAS p.G12C mutant NSCLCs (cohort A) and CRCs, PDACs, and other solid tumors (Cohort B) and have progressed after standard therapy, or standard therapy is inappropriate or unavailable.
6. Adequate organ function as defined in the below:

   Hepatic function Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 times upper limit of normal (ULN), or ≤ 5 times ULN in the presence of liver metastases. Total serum bilirubin (TBIL) ≤ 1.5 times ULN; TBIL≤3×ULN and direct bilirubin（DBIL）≤1.5×ULN in the presence of liver metastases or with Gilbert's syndrome.

   Bone marrow function No blood transfusion or hematopoietic stimulator treatment within 7 days; absolute neutrophil count (ANC) ≥1.5×10^9/L; platelets (PLT) count ≥75×10^9/L; hemoglobin (Hb) ≥ 90 g/L.

   Renal function Creatinine clearance ≥ 50 mL/min. Coagulation function International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN.
7. Female patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to the first dose. Both male and female patients of reproductive potential must be willing to abstain completely or agree to use an appropriate method of contraception during the entire study duration and for at least 3 months after the last dose of study medication.
8. Willingness and ability to give informed consent and follow protocol procedures, and comply with follow-up visit requirements.

Exclusion Criteria:

1. Dose-escalation phase: patients with known driver alterations other than KRAS p.G12C, e.g., EGFR, ALK, ROS1, RET, TRK, etc. (Enrollment of patients with co-mutations may be discussed with the investigator).
2. Dose-expansion phase: prior use of selective KRAS inhibitors.
3. Patients who received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immunotherapy, and other anti-tumor treatment within 3 weeks before the first administration, except for the following: Nitrosourea or mitomycin C was received within 6 weeks before the first administration; Oral fluoropyrimidines and small molecule targeted drugs within 2 weeks or 5 half-lives of the drug (whichever is longer) prior to the first administration; Chinese proprietary medicines with anti-tumor indications were received within 2 weeks before the first administration.
4. Received other unapproved investigational drugs or treatments within 4 weeks prior to the first administration.
5. Have undergone major organ surgery (excluding needle biopsy) or had significant trauma within 4 weeks prior to the first administration.
6. Unresolved toxicities from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade ≤ 1(exceptions for toxicities judged by the investigator to be of no safety concern, e.g. alopecia, grade 2 peripheral neurotoxicity, etc.).
7. Presence of spinal cord compression, meningeal metastases, clinically symptomatic brain metastases, or need for increased steroid doses to control central nervous system (CNS) disease; patients with symptomatic CNS metastases that are already under control may be eligible for this study.
8. Patients with active infection who need systematic anti-infective therapy within 2 weeks prior to the first administration.
9. Active hepatitis (Hepatitis B: Hepatitis B virus surface antigen [HBsAg] positive with HBV DNA ≥2000 IU/mL; Hepatitis C: Hepatitis C virus antibody positive with HCV RNA ≥1000 IU/mL), HIV antibody positive, active syphilis (double positive for syphilis non-specific and syphilis specific antibodies) that is uncontrolled by treatment and inappropriate for enrollment as determined by the investigator.
10. Presence of other lung diseases requiring systemic treatment or severe lung diseases such as active tuberculosis, interstitial lung disease, etc., which in the opinion of the investigator may affect the interpretation of the study results or place the patient at high risk;
11. A history of serious cardiovascular and cerebrovascular disease, including but not limited to severe cardiac rhythm and conduction abnormalities, such as ventricular arrhythmias and degree II-III atrioventricular block requiring clinical intervention; Longer QT interval at rest (QTc > 470 msec for women or > 450 msec for men); Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months prior to first administration; Heart failure with the New York Heart Association (NYHA) Heart function rating ≥ II or left ventricular ejection fraction (LVEF) < 50%; Clinically uncontrolled hypertension.
12. Strong inhibitor or inducer of CYP3A, P-glycoprotein inducer or inhibitor used within 1 week or 5 half-lives (whichever is longer) prior to the first administration or expected to be used during the study period.
13. Patients with malignancies other than tumors treated in this study (except malignancies that are cured and have not recurred within 2 years prior to study enrollment; completely resected basal cell and squamous cell skin cancer; completely resected carcinoma in situ of any type).
14. Severe gastrointestinal disease of clinical significance as determined by the investigator, including active ulcerative colitis, Crohn's disease, peptic ulcer disease, or previous surgical procedures that may have significantly affected drug absorption.
15. History of allergy to study drug components or adjuvants.
16. Pleural, abdominal, or pericardial effusions that are poorly controlled despite intervention (defined as effusion that has grown significantly within 2 weeks of removal and is symptomatic requiring re-puncture or other intervention).
17. Uncontrolled diabetes mellitus [fasting blood glucose ≥10 mmol/L and/or glycated hemoglobin (HbA1c) ≥8%], uncontrolled symptomatic hyperthyroidism or hypothyroidism, uncontrolled symptomatic hypercalcemia or hypocalcemia.
18. Have a coagulation disorder or bleeding tendency, including an arterial or venous thromboembolic event or any life-threatening bleeding event within 6 months prior to first administration, or have a lesion involving a major blood vessel, or have a bleeding tendency as determined by the investigator.
19. Pregnant or lactating women.
20. Presence of any condition that may increase the risks associated with the administration of the study drug or that may affect the interpretation of the study results, or poor patient compliance, or any other condition that, in the opinion of the investigator, makes the enrollment inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-limiting toxicities (DLTs) | 31 days after the first dose (single dose for 3 days and dose-escalation cycle 1 for 28 days)
  Number of participants with DLTs
Number of participants with adverse events | Up to 18 months
  Patients will be assessed for incidence and severity of adverse events (AEs) according to NCI-CTCAE v5.0 criteria

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax) for SY-5933 | Protocol-defined time points during 3 days after the first dose and cycle 1 (each cycle is 28 days)
  Defined as maximum observed plasma concentration
Pharmacokinetics (Tmax) for SY-5933 | Protocol-defined time points during 3 days after the first dose and cycle 1 (each cycle is 28 days)
  Defined as time to maximum plasma concentration
Pharmacokinetics (AUC0-t) for SY-5933 | Protocol-defined time points during 3 days after the first dose and cycle 1 (each cycle is 28 days)
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration
Pharmacokinetics (t½) for SY-5933 | Protocol-defined time points during 3 days after the first dose and cycle 1 (each cycle is 28 days)
  Defined as the apparent plasma terminal phase disposition half-life
Overall Response Rate (ORR) as assessed by RECIST 1.1 criteria | Up to 24 months
  Preliminary measure of anti-tumor activity of SY-5933 in patients with KRAS p.G12C mutant advanced tumor
Disease control rate (DCR) as assessed by RECIST 1.1 criteria | Up to 24 months
  Preliminary measure of anti-tumor activity of SY-5933 in patients with KRAS p.G12C mutant advanced tumor
Duration of response (DOR) | Up to 24 months
  Preliminary measure of anti-tumor activity of SY-5933 in patients with KRAS p.G12C mutant advanced tumor

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Sun, PhD, Study Director — Shouyao Holdings (Beijing) Co. LTD
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, China